CLINICAL TRIAL: NCT02351323
Title: Novel Type 2 Diabetes Mellitus Preventive Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-27812 (K23DK082732)
Record Dates: First submitted 2014-12-17; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine + Lifestyle change (Experimental): Glutamine 30 grams/day X 12-14 weeks, Lifestyle change
  Interventions: Drug: Glutamine (Pharmacological doses); Behavioral: Lifestyle change
- No glutamine + Lifestyle change (Placebo Comparator): Lifestyle change
  Interventions: Behavioral: Lifestyle change

INTERVENTIONS:
Drug: Glutamine (Pharmacological doses) — 30 grams/day of glutamine for 12-14 months
  Other Names: NutreStore
  Arms: Glutamine + Lifestyle change
Behavioral: Lifestyle change — Lifestyle change as recommended by Registered Dietitian

SUMMARY:
Over the past two decades, type 2 diabetes mellitus (T2DM) has emerged from relative obscurity to become one of the most serious complications of obesity in Hispanic obese populations, especially among those with a family history of T2DM. Few therapies have demonstrated long term efficacy in combating obesity and risk of T2DM in youth. Given the emerging evidence that glutamine and leucine (building blocks of protein) may affect energy partition and thus diabetes risk, and that the relationship of glutamine and diabetic risk has been further evaluated in one adult observational cohort study but data on leucine are lacking, we plan to conduct a clinical trial to determine the efficacy of glutamine to reduce insulin resistance, a diabetes risk factor.

The primary specific aim of the research plan is to conduct a randomized, double-blind, placebo controlled, clinical trial to test the efficacy of 6 months supplements of glutamine in reducing biomarkers for insulin resistance and weight gain among 56 obese Hispanic adolescents age 12-19 years with a BMI at or above the 95th percentile and a family history of T2DM. At the end of the grant period, we will have obtained preliminary data to plan pivotal clinical trials of glutamine coupled with or without lifestyle changes.

DETAILED DESCRIPTION:
Because of recruitment difficulties the design was modified several times until April 2013 when we were able to increase recruitment. The following changes were made from initial to final study design:

1. Study moved from Clinical and Translational Science Institute (CTSI) to clinical setting (Nutrition and Fitness for Life Clinic)
2. Ages eligible expanded from 12-19 years old to 12-19.9 years old
3. Ethnicity/Race expanded from Hispanic only to include all races/ethnicities
4. Patients without a past family history of T2DM were made eligible
5. Study period was shortened from 6 months to 12-14 weeks
6. Number of required visits were reduced from 5 visits to 3 visits (all of which took place during regularly scheduled clinic appointments)
7. Open labeled but still randomized
8. Those in the Glutamine arm were provided lifestyles change intervention
9. Glycosylated hemoglobin (A1C) used instead of fasting Homeostatic Model Assessment-Insulin Resistance (HOMA-IR)
10. Non-fasting blood draw rather than a fasting blood draw was instituted

ELIGIBILITY:
Inclusion Criteria:

1. BMI (k/m2) >= 95th percentile;
2. Weight 150 - 400 pounds;
3. Language: English or Spanish (The PI speaks both English and Spanish fluently).

Exclusion Criteria:

1. History of T2DM;
2. Prior or current drug treatmeant that would effect diabetes risk
3. Use of prescription strength glucocorticoids within three months before screening,
4. History of syndrome or medical disorder associated with significant obesity;
5. Serum creatinine >1.2 mg/dL;
6. Alanine transaminase (ALT) or Aspartate aminotransferase (AST) >90 international units (IU)/L (= 3 X normal limits);
7. Total bilirubin >2.5 time the upper limit of normal;
8. History of moderate to extreme physical activity, past or current pregnancy;

9 .Use of illegal/illicit drugs;

10. Unable to comply with the protocol;

11. Any other serious disease determined by the clinician as potential study risk for the patient.

12. Have kidney or liver disorders, or conditions resulting in ammonia accumulation

13. Take Lactulose

14. Are allergic to monosodium glutamate (MSG), glutamine, or Crystal Light

15. Have manic episodes (mental illness)

16. Take medications to prevent seizures

17. Take any glutamine, supplement with glutamine, hypoglycemiants, anticonvulsivant, ADHD medications, antilipidemiants, or thyroid hormone

18. Participation in a weight loss program or use of weight loss medications within six months of screening that has resulted in 5% or more weight loss

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Weight gain | 12-14 weeks

SECONDARY OUTCOMES:
Change in A1C | 12-14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carine M Lenders, MD, ScD, MS, Principal Investigator — Physician Scientist
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States